CLINICAL TRIAL: NCT00566202
Title: A Phase IIa Multicenter, Randomized, Double-blind, Double-dummy, and Placebo- and Active Controlled Study to Investigate the Safety and Efficacy of JNJ-18038683 Administered to Subjects With Major Depressive Disorder
Brief Title: A Safety and Effectiveness Study of JNJ-18038683 in Patients With Moderate to Severe Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR014617; C-2007-007 (Other: Johnson & Johnson Pharmaceutical Research & Development, L.L.C.); NCT00761293 (obsolete NCT alias)
Record Dates: First submitted 2007-11-29; First posted 2007-12-03 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; Depression; JNJ-18038683; Escitalopram
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Escitalopram; 3-(4-chlorophenyl)-1,4,5,6,7,8-hexahydro-1-(phenylmethyl)pyrazolo(3,4-d)azepine 2-hydroxy-1,2,3-propanetricarboxylate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- JNJ-18038683 (Experimental)
  Interventions: Drug: Placebo; Drug: JNJ-18038683
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: JNJ-18038683
- Escitalopram (Active Comparator)
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Placebo — Form= capsule, route= oral use. Administration once daily for 8 weeks.
  Arms: JNJ-18038683; Placebo
Drug: Escitalopram — Type= range, unit= mg, number= 10 to 20, form= capsule, route= oral use. Administration of 10 mg daily for 1 week, 20 mg daily for 6 weeks, and 10 mg daily for 1 week.
  Arms: Escitalopram
Drug: JNJ-18038683 — Type= range, unit= mg, number= 10 to 20, form= capsule, route= oral use. Administration of 10 mg daily for 1 week, 10 or 20 mg daily for 6 weeks, and placebo daily for 1 week.
  Arms: JNJ-18038683; Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of JNJ-18038683 compared to escitalopram and placebo in patients with moderate to severe depression.

DETAILED DESCRIPTION:
This study is being done to assess safety and tolerability and to explore the effectiveness of a new, experimental drug in the treatment of moderate to severe depression. Approximately 225 patients with depression will be recruited for the study. Patients who meet study criteria will need to stop taking any depression medications they are currently using. They will be randomly assigned to one of 3 treatment arms; each patient has an equal chance of receiving 20 mg JNJ-18038683, 20 mg escitalopram, or placebo. Placebo has no active drug. Escitalopram is a drug currently approved to treat depression. This is a blinded study, ie the patient, the study doctor, and the study sponsor will not know what treatment the patient receives until all patients complete the study. Patients receiving either escitalopram or JNJ-18038683 will be titrated up to their assigned dose, receiving 10 mg doses for one week prior to increasing to 20 mg. Patients who are not able to tolerate 20 mg of JNJ-18038683 will be allowed to drop down to the 10 mg dose at any time after the titration period. Patients taking 20 mg escitalopram will receive 10 mg at their final week to taper off of the drug. Patients will receive a drug blister card at each weekly visit containing drug for the upcoming week. The study doctor and the sponsor will monitor the study for the occurrence of possible side effects. In addition to a screening visit, patients will return weekly for 9 additional study visits. After completing the study, patients may resume other depression medications. Medical and psychiatric history, physical examination, blood pressure, heart rate, temperature, weight and electrocardiograms (ECGs) will be checked periodically. Blood samples will be taken for standard safety laboratory tests as well as for the measurement of the drug blood level. Questionnaires relating to depression, sleep and sexual experience will be administered throughout the study. Each day for nine weeks, patients will take orally two JNJ-18038683 tablets, active and/or placebo, and two escitalopram capsules, active and/or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with moderate to severe major depressive disorder
* Willing to use acceptable methods of birth control throughout the study and for 3 months after
* In good general health

Exclusion Criteria:

* No history or current diagnosis of other psychiatric conditions such as bipolar disorder, psychotic disorder, general anxiety disorder, anorexia, obsessive compulsive disorder, post traumatic stress disorder, antisocial personality disorder, mental retardation, pervasive developmental disorder, or cognitive disorder
* No history or presence of drug abuse
* No use of prescription medications or herbal medications other than hormone replacement therapies
* No prior history of heart disease or current significant blood, lung, kidney, liver, heart, breathing, neurologic or thyroid disorders
* No patients who are either pregnant or nursing

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2007-12; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Explore the effectiveness of JNJ-18038683 in patients with moderate to severe depression as determined by accepted clinical assessments done throughout the study. | Clinical assessments to evaluate depression will be done 8 times at weekly visits from baseline through the Week 7 visit.

SECONDARY OUTCOMES:
Explore the safety and tolerability of JNJ-18038683 in patients with moderate to severe depression by assessing adverse events, vital signs, laboratory test results, ECGs and physical exams. | Vital signs will be collected weekly throughout the study; ECGs will be collected at screening, baseline, Wks 3 and 7; Laboratory test will be collected at screening, baseline, and Wks 1,3,5,7 and 8. Adverse Events will be throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (26):
- United States (26):
  - Little Rock, Arkansas
  - Beverly Hills, California
  - Glendale, California
  - San Diego, California
  - Bradenton, Florida
  - Maitland, Florida
  - Orlando, Florida
  - Atlanta, Georgia
  - Eagle, Idaho
  - Chicago, Illinois
  - Prairie Village, Kansas
  - Topeka, Kansas
  - Baton Rouge, Louisiana
  - Shreveport, Louisiana
  - Nutley, New Jersey
  - Brooklyn, New York
  - Cedarhurst, New York
  - Fresh Meadows, New York
  - Cincinnati, Ohio
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Norristown, Pennsylvania
  - Memphis, Tennessee
  - Austin, Texas
  - Irving, Texas
  - Richmond, Virginia